CLINICAL TRIAL: NCT03297229
Title: Effectiveness of Peer Mentoring and Blood Pressure Self-monitoring for Blood Pressure Control in Vulnerable Population in Argentina. A Randomized Clinical Trial.
Brief Title: Effect of Peer Mentoring and Blood Pressure Self-monitoring on Hypertension Control.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AR-T1087-P0001
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
Keywords: Peer mentoring; Self-monitoring; Behavioral economics; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer mentoring (Experimental): Peers will be patients with hypertension that have already been adequately controlled within the last six months. They will be selected within each center by the staff of the center and invited to participate in the study.
  Interventions: Behavioral: Peer mentoring
- Self-monitoring (Experimental): Each participant will receive a blood pressure monitor. The study nurse will teach the participant on how to use the device.
  Interventions: Behavioral: Self-monitoring
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Peer mentoring — Peers will be assigned to participants according to common socio-demographic characteristics. Each peer will be assigned up to 5 participants.
  Arms: Peer mentoring
Behavioral: Self-monitoring — Along with providing patients with a BP monitor, a "commitment contract" will be signed, in which participants commit themselves to measure their blood pressure at home at least once a week during the 3 months of the intervention. Each participant will be given a form to weekly recording their blood pressure values.
  Arms: Self-monitoring

SUMMARY:
Cardiovascular diseases are increasing throughout the developing world and are the cause of almost 16.7 million deaths each year, of which 80% occur in low and middle-income countries. As more than three fourth of the global burden of cardiometabolic diseases are related to risk factors connected with lifestyles or behaviors, such as smoking, unhealthy eating, low physical activity, and harmful consumption of alcohol. This burden could be dramatically reduced by changing individual behaviors. This study is focused on interventions that are aimed to improve the adherence to treatment in cardiovascular disease (hypertension), based on a Behavioral Economics approach. Most of public policies targeted to tackle Noncommunicable diseases utilize a rational economic model of behavior.

Behavioral economics, by using insights from cognitive psychology and other social sciences, has drawn a lot of attention for its potential to increase healthy behaviors. Interventions informed by Behavioral economics principles seek to rearrange the social or physical environment in such a way to 'nudge' people towards healthier choices and behaviors. This is an individual controlled randomized trial which will be conducted to assess whether the implementation of two strategies, blood pressure self-monitoring plus signing a "contract of commitment", and peer mentoring are effective to reduce blood pressure values over a period of 3 months, compared to usual care. This randomized trial will enroll 430 patients from 10 public primary care clinics in Argentina.

ELIGIBILITY:
Inclusion Criteria:

* Adults (21 years and older) who only have public health coverage, and have high blood pressure (SBP ≥140 mmHg and / or DBP ≥90 mmHg)

Exclusion Criteria:

* Pregnant women, bed-bound, and patients who cannot give informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 3 months
  Net change in blood pressure levels from baseline to the end of follow-up in in each group.

SECONDARY OUTCOMES:
Controlled hypertension | 3 months
  Proportion of patients with controlled hypertension (Systolic blood pressure <140 mm Hg and diastolic blood pressure <90 mm Hg)
Adherence to antihypertensive medication | 3 months
  Proportion of patients who had adhered to antihypertensive medication according to the Morisky Green Scale.
Intensification of antihypertensive medication | 3 months
  Proportion of patients who increased the number of antihypertensive medications or increase the dose of their antihypertensive medication.
Visits to the clinic | 3 months
  Number of visits to the clinic over the 3 month period of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Irazola, MD, PhD, Principal Investigator — Institute for Clinical Effectiveness and Health Policy
Locations (10):
- Argentina (10):
  - Centro Asistencial Modelo Don Bosco, Quilmes, Buenos Aires
  - Policlínico Julio Méndez, Quilmes, Buenos Aires
  - UAP Illia, Vicente López, Buenos Aires
  - UAP Sargento Cabral, Vicente López, Buenos Aires
  - CAPS 1 Simeon Payba, Paso de los Libres, Corrientes Province
  - CAPS 10 Plurianual, Paso de los Libres, Corrientes Province
  - Centro de Atención Primaria de la Salud Dr. Balbastro, Corrientes
  - Centro de Atención Primaria de la Salud N°15 Illia, Corrientes
  - Centro de Salud nº 60 - El Mirador, Salta
  - Centro de Salud Santa Ana, Salta

REFERENCES:
- [Derived] Nejamis A, Chaparro M, Gibbons L, Poggio R, Moyano DL, Irazola V. Effectiveness of peer mentoring and self-monitoring to improve blood pressure control in a vulnerable population in Argentina: Pragmatic randomized open-label controlled trial. Chronic Illn. 2024 Dec;20(4):684-698. doi: 10.1177/17423953231187170. Epub 2023 Jul 11. PMID 37431737